CLINICAL TRIAL: NCT02550236
Title: Prospective Population-based Childhood Cohort Study in the Leipzig Area Investigating Genetic, Environmental, and Metabolic Factors and Their Association With the Development of Civilization Diseases
Brief Title: LIFE Child (LIFE Leipzig Research Centre for Civilization Diseases)
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: European Social Fund (Other); European Regional Development Fund (Other); Free State of Saxony (Unknown); Helmholtz Center for Environmental Research Leipzig (Unknown); Leipzig Research Center for Early Child Development (Unknown); Robert Koch Institute Berlin (Unknown)
Responsible Party: Principal Investigator, Antje Koerner, Prof. Dr. med., Prof. Dr. med. Antje Körner, University of Leipzig
Other Study IDs: LIFE Child Leipzig
Record Dates: First submitted 2014-12-15; First posted 2015-09-15 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Child Development
Keywords: Children; Pregnancy; Growth; Lifestyle; Metabolic and cardiovascular health; Birth; Development; Reference Values

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * blood samples for mRNA and DNA analysis
  * serum samples
  * plasma samples
  * serum samples from oral glucose tolerance testing
  * urine samples
  * stool samples
  * hair samples
  * mother's milk samples
  * cord blood samples
  * placenta samples
  * dental plaque samples
  * milk teeth samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LIFE Child Health: The LIFE Child HEALTH cohort is a sample of over 5.000 children and adolescents. A basic program that will be carried out annually at each study centre visit. This program includes clinical history (perinatal and past medical history, medications, allergies, immunizations, developmental history and family history) clinical examination, collection of blood, hair, stool and urine samples, anthropometry and different age-dependent questionnaires. Questionnaires are completed by the parents and starting at the age of ten years also by the child itself.
- LIFE Child Obesity: The LIFE Child OBESITY cohort is a sample of 500 obese children and adolescents that will be assessed and compared to a lean control group (N=500) with equally detailed phenotyping including metabolic and cardiovascular evaluation. The LIFE Child OBESITY cohort (including the control group) performs the basic program of the LIFE Child HEALTH cohort plus additional parameters such as electrical bioimpedance, assessment of basal metabolic rate, oral glucose tolerance test, liver elastography and spirometry.
- LIFE Child Health: Pregnancy/Birth: The LIFE child Pregnancy/Birth cohort is a sample of over 1,200 pregnant women and their offspring. Prenatal examinations are conducted during the 24th to 26th and 34th to 36th week of gestation. During the first year of life, data is collected from children at 3, 6 and 12 month of age.

SUMMARY:
The Leipzig Research Centre for Civilization Diseases (LIFE) Child Study is a prospective longitudinal population-based study with a life course approach to health and disease.

The LIFE Child Study focuses on two main research objectives:

* What are premises of normal growth, development and health in children?
* Which factors contribute to the development of non-communicable diseases such as childhood obesity and its co-morbidities, atopy and mental health problems?

Detailed assessments will be conducted alongside long-term storage of biological samples in 1,000 pregnant women and more than 5,000 children and their families.

DETAILED DESCRIPTION:
* The LIFE Child study is part of LIFE, a life sciences research program of the University of Leipzig (Leipzig Research Centre for Civilization Diseases - LIFE). The measurements are performed in a well-equipped research centre located on the premises of the University Hospital of Leipzig.
* The study collects detailed information from clinical examinations, questionnaires and interviews and includes a collection of several types of biological materials at various time points (urine, stool, hair, blood for direct analyses, genomic DNA, dried blood spots, paxgenes (for RNA isolation and expression/eQTL studies). Children and adolescents from 0 to 20 years at baseline and their families are included. Participants are followed annually over a period of several years irrespective of the age at the first participation in the study until they reach the age of 20.
* Prenatal examinations are conducted in the 24th and 36th week of gestation and postnatal examinations in the 3rd, 6th and 12th month in the offspring. The birth cohort study collects detailed information from clinical examinations, questionnaires and interviews and biological materials (blood, cord blood, placental tissue, breast milk, hair, urine and stool)
* In addition, the LIFE Child study focuses in the disease cohort LIFE Child OBESITY and disease free controls in more detail. The aim of these subgroups is to examine aetiological associations and comorbidities with more in-depth methods.

ELIGIBILITY:
Inclusion Criteria:

* children with their families and pregnant women of the area of Leipzig

Exclusion Criteria:

* severe diseases

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The LIFE Child study is a prospective longitudinal population-based cohort study. All children with their families and pregnant women of the area of Leipzig are eligible to participate in the LIFE Child study. This sample is supposed to represent the population of the city.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2010-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Civilization diseases and their risk factors | 20 years
  Assess lifestyle, metabolic and genetic risk factors of civilization diseases (e.g. diabetes mellitus, obesity, allergy, cardiovascular diseases) from fetal life to adulthood.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Körner, Prof., MD, Principal Investigator — University of Leipzig
Locations (1):
- LIFE Leipzig Research Centre for Civilization Diseases, University of Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Poulain T, Schmidt R, Kiess W, Krause S, Golz S, Meigen C. Performance on an attention test is positively related to reading but negatively related to watching TV and playing video games in children. BMC Pediatr. 2025 Oct 28;25(1):872. doi: 10.1186/s12887-025-06260-w. PMID 41146137
- [Derived] Durgen P, Wolfle PJ, Ceglarek U, Kratzsch J, Kiess W, Vogel M. New sex hormone-binding globulin and estimated free testosterone reference intervals for children and adolescents: The effects of age, sex, BMI and oral contraceptives. Clin Chim Acta. 2026 Jan 15;579:120621. doi: 10.1016/j.cca.2025.120621. Epub 2025 Sep 25. PMID 41015329
- [Derived] von Heimburg P, Baber R, Willenberg A, Wolfle P, Kratzsch J, Kiess W, Vogel M. Effect of sex, pubertal stage, body mass index, oral contraceptive use, and C-reactive protein on vitamin D binding protein reference values. Front Endocrinol (Lausanne). 2025 Feb 18;16:1470513. doi: 10.3389/fendo.2025.1470513. eCollection 2025. PMID 40041287
- [Derived] Gruning Parache L, Vogel M, Meigen C, Kiess W, Poulain T. Family structure, socioeconomic status, and mental health in childhood. Eur Child Adolesc Psychiatry. 2024 Jul;33(7):2377-2386. doi: 10.1007/s00787-023-02329-y. Epub 2023 Dec 26. PMID 38147107
- [Derived] Wex I, Geserick M, Leibert T, Igel U, Sobek C, Meigen C, Kiess W, Vogel M. Active school transport in an urban environment:prevalence and perceived barriers. BMC Public Health. 2023 Mar 23;23(1):557. doi: 10.1186/s12889-023-15464-7. PMID 36959624
- [Derived] Schild CE, Meigen C, Kappelt J, Kiess W, Poulain T. Associations between sociodemographic and behavioural parameters and child development depending on age and sex: a cross-sectional analysis. BMJ Open. 2022 Nov 2;12(11):e065936. doi: 10.1136/bmjopen-2022-065936. PMID 36323480
- [Derived] Kiess A, Green J, Willenberg A, Ceglarek U, Dahnert I, Jurkutat A, Korner A, Hiemisch A, Kiess W, Vogel M. Age-Dependent Reference Values for hs-Troponin T and NT-proBNP and Determining Factors in a Cohort of Healthy Children (The LIFE Child Study). Pediatr Cardiol. 2022 Jun;43(5):1071-1083. doi: 10.1007/s00246-022-02827-x. Epub 2022 Mar 12. PMID 35277733
- [Derived] Hovestadt I, Kiess W, Lewien C, Willenberg A, Poulain T, Meigen C, Korner A, Vogel M. HbA1c percentiles and the association between BMI, age, gender, puberty, and HbA1c levels in healthy German children and adolescents. Pediatr Diabetes. 2022 Mar;23(2):194-202. doi: 10.1111/pedi.13297. Epub 2021 Dec 20. PMID 34877761
- [Derived] Menzel P, Vogel M, Austin S, Sprenger N, Grafe N, Hilbert C, Jurkutat A, Kiess W, Binia A. Concentrations of oligosaccharides in human milk and child growth. BMC Pediatr. 2021 Oct 30;21(1):481. doi: 10.1186/s12887-021-02953-0. PMID 34717578
- [Derived] Ziegelasch N, Vogel M, Korner A, Koch E, Jurkutat A, Ceglarek U, Dittrich K, Kiess W. Cystatin C relates to metabolism in healthy, pubertal adolescents. Pediatr Nephrol. 2022 Feb;37(2):423-432. doi: 10.1007/s00467-021-05209-2. Epub 2021 Aug 25. PMID 34432142
- [Derived] Surup H, Vogel M, Koerner A, Hiemisch A, Oelkers L, Willenberg A, Kiess W, Kratzsch J. Pediatric Reference Intervals for Thyrotropin, Free Triiodothyronine, and Free Thyroxine and the Relevance of Body Mass Index and Puberty in Measurement Interpretation. Thyroid. 2021 Aug;31(8):1192-1202. doi: 10.1089/thy.2020.0780. Epub 2021 Jun 21. PMID 33906420
- [Derived] Michel L, Shevlyakova M, Ni Cleirigh E, Eckhardt E, Holvoet S, Nutten S, Sprenger N, Korner A, Vogel M, Nembrini C, Kiess W, Blanchard C. Novel approach to visualize the inter-dependencies between maternal sensitization, breast milk immune components and human milk oligosaccharides in the LIFE Child cohort. PLoS One. 2020 Apr 21;15(4):e0230472. doi: 10.1371/journal.pone.0230472. eCollection 2020. PMID 32315306
- [Derived] Dathan-Stumpf A, Vogel M, Jank A, Thiery J, Kiess W, Stepan H. Reference intervals of serum lipids in the second and third trimesters of pregnancy in a Caucasian cohort: the LIFE Child study. Arch Gynecol Obstet. 2019 Dec;300(6):1531-1539. doi: 10.1007/s00404-019-05342-2. Epub 2019 Oct 30. PMID 31667609
- [Derived] Haas M, Hiemisch A, Vogel M, Wagner O, Kiess W, Poulain T. Sensation seeking in 3- to 6-year-old children: associations with socio-demographic parameters and behavioural difficulties. BMC Pediatr. 2019 Mar 11;19(1):77. doi: 10.1186/s12887-019-1450-6. PMID 30857528
- [Derived] Ziegelasch N, Vogel M, Muller E, Tremel N, Jurkutat A, Loffler M, Terliesner N, Thiery J, Willenberg A, Kiess W, Dittrich K. Cystatin C serum levels in healthy children are related to age, gender, and pubertal stage. Pediatr Nephrol. 2019 Mar;34(3):449-457. doi: 10.1007/s00467-018-4087-z. Epub 2018 Nov 20. PMID 30460495
- [Derived] Poulain T, Peschel T, Vogel M, Jurkutat A, Kiess W. Cross-sectional and longitudinal associations of screen time and physical activity with school performance at different types of secondary school. BMC Public Health. 2018 Apr 27;18(1):563. doi: 10.1186/s12889-018-5489-3. PMID 29703168
- [Derived] Rieger K, Vogel M, Engel C, Ceglarek U, Harms K, Wurst U, Lengfeld H, Richter M, Kiess W. Does physiological distribution of blood parameters in children depend on socioeconomic status? Results of a German cross-sectional study. BMJ Open. 2018 Mar 1;8(3):e019143. doi: 10.1136/bmjopen-2017-019143. PMID 29500207
- See also: List of all publications, sorted by topic — https://home.uni-leipzig.de/lifechild/publications/